CLINICAL TRIAL: NCT02874235
Title: Music Therapy Versus Treatment as Usual: A Randomized Non-inferiority Study With Traumatized Refugees Diagnosed With PTSD
Brief Title: Music Therapy and Treatment as Usual
Acronym: RCT-KTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: Det Obelske Familiefond (Unknown); Aalborg University (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-529
Record Dates: First submitted 2016-06-28; First posted 2016-08-22 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: External psychologist performs primary outcome measurement not knowing participants treatment
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy treatment (Experimental): 35 patients receiving each 16 sessions of Receptive music therapy
  Interventions: Behavioral: Receptive music therapy
- Standard treatment (Active Comparator): 35 patients receiving each 16 sessions of Psychological treatment
  Interventions: Behavioral: Psychological treatment

INTERVENTIONS:
Behavioral: Receptive music therapy — 16 sessions of a length of one hour comprising of receptive music psychotherapy with 5 - 15 minutes of music listening included
  Other Names: Modified Guided Imagery and Music
  Arms: Music therapy treatment
Behavioral: Psychological treatment — 16 sessions of a length of one hour comprising of verbal based psychotherapy based on principles from Narrative Exposure Therapy or Cognitive Behavioral Therapies
  Arms: Standard treatment

SUMMARY:
This study compares music therapy with verbal psychotherapy (treatment as usual) in an outpatient psychiatric clinic for traumatized refugees. Based on positive results from a pilot study, the randomized clinical trial has a non-inferiority design to detect whether music therapy is not less effective than verbal therapy carried out by psychologists and can serve as a complementary treatment modality (n=70).

The participants are adult Arabic, English or Danish speaking refugees suffering from posttraumatic stress disorder (PTSD). The patients are referred to outpatient treatment by their medical doctor. Data collection takes place in three locations of the clinic in Region Zealand, Denmark. The music therapy method used is Guided Imagery and Music (GIM).

Primary outcome is pre, post and 6 months follow-up measures of HTQ (Harvard Trauma Questionaire) and two measures of PTSD-8 during treatment. Secondary outcomes are pre, post and 6 months follow-up measures of Quality of Life Questionnaire (WHO-5), Dissociation Symptom Scale (DSS), Somatoform Dissociation Questionaire (SDQ-20), Revised Adult Attachment Scale (RAAS) and physiological measures (salivary oxytocin, betaendorphin and Substance P).

DETAILED DESCRIPTION:
Subjects are randomized to 16 sessions of trauma modified GIM or 16 sessions of verbal psychotherapy (standard treatment).

N (70) is based on a power calculation using HTQ measures from similar refugee studies, with an estimated effect size in the range 0.6-0.8.

Sampling All baseline measures are scored during interview with a therapist before randomization. The primary post and follow-up measures (HTQ-R) are scored during interviews conducted by external psychologists blinded to the treatment group. The secondary post and follow-up measures are self-report questionnaires scored by the patients with the help of an educated translator who is blinded with regards to the treatment group.

0.5 ml salivary samples are collected in plastic tubes and stored at -20 degrees C.

The concentration of tree hormones (oxytocin, betaendorphin, substance P) are analyzed in a multiplex solution.

Intervention

The intervention is a phased trauma-oriented modification (tmGIM) of the Bonny Method of Guided Imagery and Music (GIM), where music listening and spontaneous imagery in an altered state of consciousness is used within a psychotherapeutic session to promote inner transformation and growth. The method was adapted by certain constraints:

Using only a limited selection of music with musical parameters, that fully support the trauma-oriented therapeutic goals and do not provoke flashbacks.

Using short music listening periods (2-10 minutes). Listening in an upright position. Inclusion of music from Middle-Eastern cultures. Inclusion of psychoeducation and introductory mindfulness based exercises such as mindful breathing and body awareness. Initial focus on inner resources such as positive memories, imagining a safe place and the use of the music breathing technics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Statistical Manual of Mental Disorders (DSM-5): Posttraumatic Stress Disorder Reaction: 309.81
* Refugee status: Inhabitant in Denmark
* International Classification of Diseases (ICD-10): F43.1: PTSD or
* International Classification of Diseases (ICD-10): F62.0 Enduring personality change after catastrophic experience
* Referred from a general practitioner or other unit of psychiatry

Exclusion Criteria:

* International Classification of Diseases (ICD-10): F20-29 Schizophrenia or schizophrenia like diagnoses
* Active Substance Abuse
* Major Depression in connection with psychoses or suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in HTQ-R | 6 months
  DSM IV PTSD symptoms part (first 16 items) of section 4 of HTQ. the Harvard Trauma Questionnaire is a 4 point Likert scale. Scored during an interview with an external psychologist blinded to the treatment group. Measured at baseline, post-treatment and at 6 months follow up.
Change in PTSD-8 | 6 months
  DSM IV PTSD symptoms (8 of the first 16 items) of section 4 of HTQ. The Harvard Trauma Questionnaire is a Likert 4 point scale. PTSD is scored by the patient two times during treatment before session 4 and 12. This measure is also a part of the HTQ-R (Outcome 1)

SECONDARY OUTCOMES:
Change in WHO-5 | 6 months
  WHO-5 Quality of Life Scale, self-report questionnaire. Measured at baseline, post-treatment and at 6 months follow up.
Change in RAAS | 6 months
  Revised Adult Attachment Scale. Attachment in close relationship self-report questionnaire. Measured at baseline, post-treatment and at 6 months follow up.
Change in DSS | 6 months
  Dissociation Symptom Scale, self-report questionnaire. Measured at baseline, post-treatment and at 6 months follow up.
Change in SDQ-20 | 6 months
  Somatoform Dissociation Questionnaire, self-report questionnaire. Measured at baseline, post-treatment and at 6 months follow up.
Change in Oxytocin | 6 months
  Oxytocin collected in saliva. Measured at baseline, post-treatment and at 6 months follow up and. pre- and post session in the third or fourth session and second or third last session.
Change in Beta-endorphin | 6 months
  Beta-endorphin collected in saliva. Measured at baseline, post-treatment and at 6 months follow up and pre- and post session in the third or fourth session and second or third last session.
Change in Substance P | 6 months
  Substance P collected in saliva. Measured at baseline, post-treatment and at 6 months follow up and pre- and post session in the third or fourth session and second or third last session.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Moe, Ph.D., Study Director — Research Unit, Region Zealand Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alanne, S. (2010). Music Psychotherapy with Refugee Survivors of Torture: Interpretations of Three Clinical Case Studies. Sibelius Academy.
- [Background] Alluri V, Toiviainen P, Jaaskelainen IP, Glerean E, Sams M, Brattico E. Large-scale brain networks emerge from dynamic processing of musical timbre, key and rhythm. Neuroimage. 2012 Feb 15;59(4):3677-89. doi: 10.1016/j.neuroimage.2011.11.019. Epub 2011 Nov 12. PMID 22116038
- [Background] Beck, B. D., & Mumm, H. (2015). Forskning i musikterapi - posttraumatisk stressbelastning (PTSD). Dansk Musikterapi, 12(1). Retrieved from http://vbn.aau.dk/en/publications/forskning-i-musikterapi--posttraumatisk-stressbelastning-ptsd(9a7b99e6-ce28-451e-aad3-b0dbb63fff07).html
- [Background] Blake, R. L., & Bishop, S. R. (1994). The Bonny Method of Guided Imagery and Music (GIM) in the Treatment of Post-Traumatic Stress Disorder (PTSD) with Adults in the Psychiatric Setting. Music Therapy Perspectives, 12(2), 125-129. http://doi.org/10.1093/mtp/12.2.125
- [Background] Koelsch S. Towards a neural basis of music-evoked emotions. Trends Cogn Sci. 2010 Mar;14(3):131-7. doi: 10.1016/j.tics.2010.01.002. Epub 2010 Feb 10. PMID 20153242
- [Background] Herholz SC, Halpern AR, Zatorre RJ. Neuronal correlates of perception, imagery, and memory for familiar tunes. J Cogn Neurosci. 2012 Jun;24(6):1382-97. doi: 10.1162/jocn_a_00216. Epub 2012 Feb 23. PMID 22360595
- [Background] Bruscia, K. E. (2002). Guided Imagery and Music: The Bonny Method and Beyond. Barcelona Publishers.
- [Background] Bonny, H. L. (2002). Music Consciousness: The Evolution of Guided Imagery and Music. (L. Summer, Ed.). Gilsum, NH: Barcelona Publishers.
- [Background] Körlin, D., Nybäck, H., & Goldberg, F. S. (2000). Creative arts groups in psychiatric care Development and evaluation of a therapeutic alternative. Nordic Journal of Psychiatry, 54(5), 333-340.
- [Background] Kraus N, Zatorre RJ, Strait DL. Editors' introduction to Hearing Research special issue: music: a window into the hearing brain. Hear Res. 2014 Feb;308:1. doi: 10.1016/j.heares.2013.09.013. No abstract available. PMID 24571003
- [Background] Maack, C. (2012). Outcomes and Processes of the Bonny Method of Guided Imagery and Music (GIM) and its Adaptations and Psychodynamic Imaginative Trauma Therapy (PITT) for Women with Complex PTSD. Aalborg University Denmark 2012. Retrieved from http://gim-therapie.de/Thesis.pdf
- [Background] Moe, T. (2001). Restituerende faktorer i gruppemusikterapi med psykiatriske patienter - baseret på en modifikation af Guided imagery and Music (GIM) (PhD Thesis). Aalborg University Denmark. Retrieved from http://www.wfmt.info/Musictherapyworld/modules/archive/dissertations/pdfs/TorbenM.pdf